CLINICAL TRIAL: NCT05342350
Title: Surveillance and Treatment Of Primary Hepatocellular Carcinoma: An International Cohort Study of High-Risk Patients for HCC Using Liquid Biopsy
Brief Title: International Study of High-Risk Patients for Hepatocellular Carcinoma Using Liquid Biopsy
Acronym: STOP-HCC
Status: Terminated | Type: Observational
Why Stopped: PI moving on from current institution
Sponsor: Johns Hopkins University (Other)
Collaborators: King Faisal Specialist Hospital & Research Center (Other); Medic Medical Center (Viet Nam) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00250209
Record Dates: First submitted 2022-04-16; First posted 2022-04-22 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Liver Cancer; Liver Cirrhosis; Hepatocellular Carcinoma; Early Stage Liver Cancer
Keywords: Early detection of liver cancer; GALAD; Liver cancer; Viet Nam; Saudi Arabia; Liver cirrhosis
MeSH Terms: conditions — Liver Neoplasms; Liver Cirrhosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: GALAD Score — GALAD score, a blood-based biomarker panel (gender, age, AFP, AFP-L3%, DCP)

SUMMARY:
This study has two purposes. One is to conduct a phase IV biomarker validation study in which the investigators will prospectively survey a cohort of patients at risk for liver cancer using semi-annual abdominal ultrasound and GALAD Score for 5 years. The GALAD score is a serum biomarker-based panel that can aid in early detection among patients with a high risk for liver cancer. One is to establish a bio-repository of longitudinally collected bio-specimens from patients with fibrosis/cirrhosis as a reference set for future research.

DETAILED DESCRIPTION:
Vietnam and Saudi Arabia have some of the highest disease burdens of liver cancer globally. Early detection in asymptomatic patients who are at risk for liver is a strategy to improve survival outcomes in liver cancer management. GALAD score (gender, age, alpha-feto protein (AFP)-L%, AFP and DCP) is a serum biomarker-based panel that can improve HCC early detection in patients with liver fibrosis and cirrhosis. In case-control studies and studies with the design of prospective specimen collection, and retrospective blinded evaluation, GALAD has demonstrated promising clinical utility. However, in order to ascertain its potential role in the surveillance of liver cancer early detection, GALAD needs to be validated prospectively for clinical surveillance of liver cancer (i.e. phase IV biomarker validation study). Thus, the investigators propose to conduct a phase IV biomarker validation study to prospectively survey a cohort of patients at risk for HCC (i.e. patients with compensated cirrhosis and irrespective of cirrhosis etiologies), using semi-annual abdominal ultrasound and GALAD Score for 5 years. In doing so, the investigators aim to validate the potential role of GALAD Score for clinical surveillance and early detection of HCC in Vietnam and Saudi Arabia. Additionally, the investigators will collect and archive biospecimens to develop a bio-repository for liver disease. The biorepository will encourage the sharing of biospecimens and collaboration among physicians or physician-researchers between the US, Vietnam, and Saudi Arabia.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study and up to 5 years post-study follow up
3. Adults aged 18 or older
4. Both genders and all ethnicities
5. Willingness to give written, informed consent to be enrolled into the database
6. Collection of biosamples (serum, plasma, and urine) at each of the 6 months follow up during the study duration
7. Individuals already confirmed to have cirrhosis with MELD ≤ 15 from any etiology (chronic HBV, chronic HCV, NASH cirrhosis, etc.)
8. For chronic HBV and/or /HCV carrier, with or without on treatment
9. Reside in Vietnam or Saudi Arabia at the time of study and provides contact information (email and/or cell phone number for texting)
10. No prior or current treatment of HCC
11. No cancer history within 5 years
12. No participation in a trial for HCC Treatment
13. No prior solid organ transplant
14. Albumin, Bilirubin, Creatinine and INR labs within past 30 days
15. Imaging showing no HCC within 180 days
16. Diagnosis of fibrosis and cirrhosis based on: histology, image showing cirrhotic liver with splenomegaly and platelets <120 mm3, or esophageal or gastric varices on endoscopy AND presence of chronic liver disease/Fibroscan/Fib-4/APRI/ARFI. For viral hepatitis, kPa>=9kPa, APRI >=1; for NAFLD/NASH (FIB-4 > 1.3 & TE > 8kPa)
17. No significant hepatic decompensation
18. No hepatorenal syndrome
19. AFP labs within 180 days irrespective of AFP titer
20. Two phone numbers and personal identification numbers (CMND number)
21. No known AIDS related diseases
22. No significant co-morbid conditions with life expectancy <5 years
23. No other cancer(s)

Exclusion Criteria:

1. Decompensated cirrhosis (variceal bleeding, hepatic encephalopathy, ascites, spontaneous bacterial peritonitis, and/or hepatorenal syndrome) or MELD>15
2. Individuals who already have HCC, with or without HCC treatment
3. On liver transplantation list or anticipated to be on the liver transplantation list during the study duration
4. Individuals who cannot, do not want to, or refused to sign the informed consent form (ICF)
5. Any serious or active medical or psychiatric illness, which, in the opinion of the investigator, would interfere with patient treatment, assessment or compliance with the protocol
6. Documentation was not adequate
7. Taking Vitamin K within 7 days prior to clinic follow or having disease affecting Vitamin K levels.
8. Known HIV positive
9. Active drug use or dependence that, in the opinion of the study investigator, would interfere with adherence to study requirements

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Persons with compensated cirrhosis (e.g. MELD 15 or lower)
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-06-07 (Actual); Study Completion 2025-06-07 (Actual)

PRIMARY OUTCOMES:
GALAD performance for liver cancer early detection | 5 years
  Performance of GALAD score determined in association with liver cancer detection by LiRADS criteria in a cohort with compensated cirrhosis undergoing prospective surveillance every 6 months for 5 years.

SECONDARY OUTCOMES:
Establishment of a bio-repository of longitudinally collected from patients with cirrhosis to be used for future studies | 5 years
  Proportion of study participants agrees to consent for bio-specimen when invited

CONTACTS AND LOCATIONS:
Overall Officials: Doan Dao, MD, Principal Investigator — Johns Hopkins University
Locations (10):
- Saudi Arabia (5):
  - King Faisal Specialist Hospital and Research Center in Jeddah, Jeddah
  - National Guard Hospital in Jeddah, Jeddah
  - King Faisal Specialist Hospital and Research Centre in Riyadh, Riyadh
  - King Saud University Medical Center, Riyadh
  - National Guard Hospital in Riyadh, Riyadh
- Vietnam (5):
  - Binh An Hospital, Rach Gia, Kien Giang
  - Medic Ca Mau, Cà Mau
  - Dong Da Hospital, Hà Nội
  - Institute of Gastroenterology and Hepatology, Hà Nội
  - Medic Medical Center-Ho Chi Minh City, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Truong TN, Pham TND, Hoang LB, Nguyen VT, Dao HV, Dao DVB, Alessy S, Pham HB, Pham TTT, Nguyen LDD, Nguyen K, Abaalkhail F, Manal M, Mawardi M, AlZahrani M, Alswat K, Alghamdi H, Sanai FM, Siddiqui MA, Nguyen NH, Vaidya D, Phan HT, Johnson PJ, Alqahtani SA, Dao DY. Surveillance and treatment of primary hepatocellular carcinoma (aka. STOP HCC): protocol for a prospective cohort study of high-risk patients for HCC using GALAD-score. BMC Cancer. 2023 Sep 18;23(1):875. doi: 10.1186/s12885-023-11167-9. PMID 37723439